CLINICAL TRIAL: NCT03569332
Title: Effect of the Mobile Self-input Tool of Incentive Spirometer on Its Usage by Patients : a Randomized Clinical Trial
Brief Title: Effect of the Mobile Self-input Tool of Incentive Spirometer (RCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-02-135
Record Dates: First submitted 2018-05-25; First posted 2018-06-26 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Gastrectomy
Keywords: Incentive Spirometer
MeSH Terms: interventions — Clinical Alarms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Participants will receive the mobile self-input tool providing alarm on tablet, and their practicing rate will be sent to Nurse's Dashboard.
  Interventions: Other: Alarm; Other: Nurse's dashboard
- Control Group (No Intervention): Participants will receive the mobile self-input tool on tablet (to compare the rate with Test group). But it won't contain alarm function and their practicing rate won't be sent to Nurse's Dashboard, either.

INTERVENTIONS:
Other: Alarm — 1. Alarm is provided from 9am to 9pm.
  2. Alarm is active every 50 minutes if the exercise goal(10 times/hour) hasn't satisfied.
  Arms: Test Group
Other: Nurse's dashboard — 1. Wireless data transmission system
  2. The practicing rate of participants on study group is sent to Nurse's Dashboard.
  3. It is only to display.
  Arms: Test Group

SUMMARY:
This study evaluates the effectiveness of the mobile self-input tool providing alarm and visual motivation, how much more it can encourage practicing of incentive spirometer undergoing post-operative patients under general anesthesia. Half of participants will receive the mobile self-input tool providing alarm, and their practicing rate will be sent to Nurse's Dashboard. While the other half will receive the mobile self-input tool, but it won't contain alarm function and their practicing rate won't be sent to Nurse's Dashboard, either.

DETAILED DESCRIPTION:
1. Background : Active respiratory therapy like incentive spirometer is needed to prevent pulmonary complications for patients undergoing post-operative under general anesthesia. But in many cases, patients don't practicing it for their pain, or they just forget doing it. And medical staffs are having difficulties in checking how well the patients follow the directions for doing incentive spirometer. Insufficient practicing incentive spirometer and deep breathing cause delay their health recovery.

   Therefore, we want to make some tools which can encourage the patients' practicing for incentive spirometer and also supply the objective achievement of patients to medical staffs.
2. Objective : This study evaluates the effectiveness of the mobile self-input tool providing alarm and visual motivation, how much more it can encourage practicing of incentive spirometer undergoing post-operative patients under general anesthesia.
3. Design: RCT (randomized controlled trial)
4. Setting: In the Department of Gastrointestinal Surgery at the Samsung Medical Center
5. Enrollment : 44 patients undergoing gastrectomy.
6. Intervention 6-1) For study group : participants on study group are received self-input tool with alarm system on tablet.

   Alarm is provided only if insufficient practice (less than 10 times/hour) from 9am to 9pm. The practicing rate is sent to Nurse's Dashboard.

   6-2) For control group : participants on control group are received self-input tool without alarm on tablet. Their practicing rate is not sent to Nurse's Dashboard.
7. Scoring by practicing incentive spirometer from 9 am to 9 pm. (Only when a subject practiced more than 10 times per hour, the subject get 10 points) (Full score 240)
8. Study period : for 48hrs from one day to 3rd day after patient's operation
9. Satisfaction survey (SUS) after study(3rd day after operation)

ELIGIBILITY:
Inclusion Criteria:

* A subject undergoing total gastrectomy or subtotal gastrectomy by robotic surgery, laparoscopic surgery or open surgery
* A subject who got surgery under general anesthesia
* A Subject receiving a prescription of using incentive spirometer
* A subject who voluntarily agrees and signs

Exclusion Criteria:

* Disorientation
* Unscheduled emergency surgery
* a subject who has difficulty in active breathing exercise due to problems such as heart disease, brain disease, chronic lung disease, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Total number of practicing incentive spirometer that subjects input by themselves on the mobile self-input tool and scoring by practicing incentive spirometer from 9 am to 9 pm. | Only collecting the numbers of practicing between 9 am and 9 pm for two days, from 1st day to 3rd day after operation.
  Only when a subject practiced more than 10 times per hour, the subject get 10 points

SECONDARY OUTCOMES:
Collecting subject's medical records related to pulmonary complication | From one day after subject's operation to the date the subject leaves(discharges) the hospital. (Average duration is for 4~5days)
  such as body temperature, laboratory results and Chest X-ray.
Satisfaction Survey for mobile self-input tool | 3rd day after operation
  Scoring by the answers of the Questionnaire of Satisfaction (SUS)

CONTACTS AND LOCATIONS:
Overall Officials: Wonchul Cha, Doctoral, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gangnam, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Soh JY, Lee SU, Lee I, Yoon KS, Song C, Kim NH, Sohn TS, Bae JM, Chang DK, Cha WC. A Mobile Phone-Based Self-Monitoring Tool for Perioperative Gastric Cancer Patients With Incentive Spirometer: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Feb 19;7(2):e12204. doi: 10.2196/12204. PMID 30777844